CLINICAL TRIAL: NCT01164137
Title: Eliminating Risk of Preventable Adverse Drug Events at the Hospital-community Interface of Care: to Develop and Test a Community-based Medication Reconciliation Program and a Risk Prediction Model That Identifies High-risk Patient Groups
Brief Title: Eliminating Risk of Preventable Adverse Drug Events at the Hospital-community Interface of Care
Acronym: CMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Westview Physician Collaborative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CMPA#2026
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Adverse Drug Events
Keywords: Adverse Drug Events; Medication Reconciliation; Pharmacist-led Intervention
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Medication Reconciliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medication Reconciliation Intervention (Experimental): Participants receiving a pharmacist-led home intervention conducted within 72 hours of hospital discharge aimed at identifying and correcting medication discrepancies.
  Interventions: Behavioral: Medication Reconciliation
- Medication Reconciliation Non-Interven. (No Intervention): Participants not receiving a pharmacist-led home intervention conducted within 72 hours of hospital discharge aimed at identifying and correcting medication discrepancies.

INTERVENTIONS:
Behavioral: Medication Reconciliation — A pharmacist-led home intervention conducted within 72 hours of hospital discharge aimed at correcting and identifying medication discrepancies.
  Arms: Medication Reconciliation Intervention

SUMMARY:
This initiative aims to decrease the risk of medication errors at the hospital-community interface as well as health system utilization following hospital discharge by implementing a pharmacist-led medication reconciliation in the patients' home within 72 hours of hospital discharge.

DETAILED DESCRIPTION:
The goals of this initiative are to decrease the risk for medication errors at the hospital community interface of care, thus decreasing preventable adverse drug events and preventable drug-related health system utilization following hospital discharge. This initiative has four objectives that aim to:

1. Develop and test a community-based medication reconciliation process/intervention.
2. Design and conduct a randomized controlled trial to examine the impact of the intervention on post-discharge health services utilization by comparing a set of outcome variables between intervention and non-intervention groups.
3. Design a risk prediction model that helps identify patients discharged from in-patient care with the highest level of need for the intervention.
4. Determine whether a community-based medication reconciliation process/intervention adds risk reduction value to individuals who have undergone an in-hospital medication reconciliation.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the WestView Health Centre Medicine/Family Health Unit with at least one medication at discharge.

Exclusion Criteria:

* First Nations persons
* Residents of continuing care or assisted living facilities
* Persons not residing in the Edmonton, AB, Canada region
* Persons who obtain a score of 19 or less on the Mini Mental State Examination (MMSE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2008-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Bailey, M.D., Principal Investigator — Westview Physician Collaborative; Grace Moe, M.Sc.P.T., Study Director — WestView Primary Care Network
Locations (1):
- WestView Health Centre, Stony Plain, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period began November 1, 2008 and ended June 30, 2010.
Pre-assignment Details: Three participants were excluded from the trail before assignment to groups because they obtained a score of 19 or less on the Mini Mental State Examination (MMSE).
Groups:
- Experimental: Medication Reconciliation Intervention: Medication Reconciliation : Participants receiving a pharmacist-led home intervention conducted within 72 hours of hospital discharge aimed at correcting and identifying medication discrepancies.
- Control: Medication Reconciliation Non-Intervention: Medication Reconciliation : Participants not receiving a pharmacist-led home intervention conducted within 72 hours of hospital discharge aimed at correcting and identifying medication discrepancies.
Period: Overall Study
Arm/Group | Experimental: Medication Reconciliation Intervention | Control: Medication Reconciliation Non-Intervention
Started | 80 | 76
Completed | 77 | 76
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Medication Reconciliation Intervention | Control: Medication Reconciliation Non-Intervention | Total
Number analyzed (Participants) | 80 | 76 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 16 | 50
  >=65 years | 46 | 60 | 106
Age Continuous [Mean (Standard Deviation); unit: years] | 68.40 (14.70) | 72.59 (13.27) | 70.48 (14.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 33 | 74
  Male | 39 | 43 | 82
Region of Enrollment [Number; unit: participants]
  Canada | 80 | 76 | 156

OUTCOME MEASURES:

1. Primary Outcome: Health Services Utilization 3 Months Following Hospital Discharge
Description: Mean health services utilization 3 months following hospital discharge. The specific health services utilization was re-admission to hospital, admission to home care, admission to long-term care and visits to emergency departments.
Time Frame: 3 Months
Measure: Mean (Standard Error); unit: Health Services Utilizations
Arm/Group | Experimental: Medication Reconciliation Intervention | Control: Medication Reconciliation Non-Intervention
Number analyzed (Participants) | 77 | 76
Health Services Utilizations | 3.33 (.35) | 3.40 (.29)
Statistical Analysis 1: Comparison: Experimental: Medication Reconciliation Intervention vs Control: Medication Reconciliation Non-Intervention; Test type: Superiority or Other; p = .87, t-test, 2 sided; Mean Difference (Final Values) = -.07, 95% CI 2-sided [-.98 to .84]

2. Primary Outcome: Health Services Utilization 6 Months Following Hospital Discharge
Description: Mean health services utilization 6 months following hospital discharge. The specific health services utilization was re-admission to hospital, admission to home care, admission to long-term care and visits to emergency departments.
Time Frame: 6 Months
Measure: Mean (Standard Error); unit: Health Services Utilizations
Arm/Group | Experimental: Medication Reconciliation Intervention | Control: Medication Reconciliation Non-Intervention
Number analyzed (Participants) | 77 | 76
Health Services Utilizations | 4.57 (.52) | 3.93 (.35)
Statistical Analysis 1: Comparison: Experimental: Medication Reconciliation Intervention vs Control: Medication Reconciliation Non-Intervention; Test type: Superiority or Other; p = .32, t-test, 2 sided; Mean Difference (Final Values) = .63, 95% CI 2-sided [-.62 to 1.88]

3. Primary Outcome: Health Services Utilization 9 Months Following Hospital Discharge
Description: Mean health services utilization 9 months following hospital discharge. The specific health services utilization was re-admission to hospital, admission to home care, admission to long-term care and visits to emergency departments.
Time Frame: 9 Months
Measure: Mean (Standard Error); unit: Health Services Utilizations
Arm/Group | Experimental: Medication Reconciliation Intervention | Control: Medication Reconciliation Non-Intervention
Number analyzed (Participants) | 77 | 76
Health Services Utilizations | 5.71 (.80) | 4.49 (.41)
Statistical Analysis 1: Comparison: Experimental: Medication Reconciliation Intervention vs Control: Medication Reconciliation Non-Intervention; Test type: Superiority or Other; p = .18, t-test, 2 sided; Mean Difference (Final Values) = 1.21, 95% CI 2-sided [-.57 to 3.01]

4. Primary Outcome: Health Services Utilization 12 Months Following Hospital Discharge
Description: Mean health services utilization 12 months following hospital discharge. The specific health services utilization was re-admission to hospital, admission to home care, admission to long-term care and visits to emergency departments.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: Health Services Utilizations
Arm/Group | Experimental: Medication Reconciliation Intervention | Control: Medication Reconciliation Non-Intervention
Number analyzed (Participants) | 77 | 76
Health Services Utilizations | 6.74 (.94) | 5.03 (.48)
Statistical Analysis 1: Comparison: Experimental: Medication Reconciliation Intervention vs Control: Medication Reconciliation Non-Intervention; Test type: Superiority or Other; p = .11, t-test, 2 sided; Mean Difference (Final Values) = 1.71, 95% CI 2-sided [-.39 to 3.81]

5. Primary Outcome: Health Services Utilization 18 Months Following Hospital Discharge
Description: Mean health services utilization 18 months following hospital discharge. The specific health services utilization was re-admission to hospital, admission to home care, admission to long-term care and visits to emergency departments.
Time Frame: 18 months
Measure: Mean (Standard Error); unit: Health Services Utilizations
Arm/Group | Experimental: Medication Reconciliation Intervention | Control: Medication Reconciliation Non-Intervention
Number analyzed (Participants) | 77 | 76
Health Services Utilizations | 7.80 (1.06) | 5.95 (.59)
Statistical Analysis 1: Comparison: Experimental: Medication Reconciliation Intervention vs Control: Medication Reconciliation Non-Intervention; Test type: Superiority or Other; p = .13, t-test, 2 sided; Mean Difference (Final Values) = 1.85, 95% CI 2-sided [-.56 to 4.27]

ADVERSE EVENTS:
Time Frame: 1 year, 7 months (i.e., November 1, 2008 to June 30, 2010)
Arm/Group | Experimental: Medication Reconciliation Intervention | Control: Medication Reconciliation Non-Intervention
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/76
Other Adverse Events (participants affected / at risk) | 0/80 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No